CLINICAL TRIAL: NCT05437354
Title: Oncologists' Thoughts and Expectations Regarding Their Patients. An Online Survey
Brief Title: Online Survey: Oncologists' Thoughts Regarding Their Patients
Acronym: OncoSurvey
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Riham H. AbdelAziz, Clinical Oncology Lecturer and consultant, Cairo University
Other Study IDs: OncoSurvey2
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Oncology
Keywords: Oncologists, Survey, Expectations
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Oncology medical staff should respond to a survey

SUMMARY:
Our study is a questionnaire targeting the medical staff in Oncology. It aims at exploring the thoughts and expectations of the medical staff in Oncology regarding their patients management and prognosis worldwide. It also investigates the factors that affect these thoughts and expectations and their effects.

DETAILED DESCRIPTION:
Oncology patients need to trust the medical staff dealing with them. They are expecting knowledge, well communication, competence .. etc. This Questionnaire is for research purpose aiming at exploring the thoughts and expectations of the medical staff in Oncology regarding their patients management and prognosis worldwide. It investigates the factors that affect these thoughts and expectations and their effects. The results of this survey will shed the light on the oncologists' side of their relationship with their patients, which is often ignored or down played.

ELIGIBILITY:
Inclusion Criteria:

1. Medical/Clinical/Radiation Oncology Physicians
2. Surgical Oncology Physicians
3. Oncology nurses

Exclusion Criteria:

* Medical staff not related to oncology field

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any Medical staff in Oncology Field worldwide, with no age limit
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
What are the most and least important factors the oncologists usually consider when they build their management plan? | Two months
  We would like to know the factors that the oncologists usually consider for a patient's management plan. This will be done via a questionnaire.

SECONDARY OUTCOMES:
How often do oncologists inform patients of the detailed management plan? and Why? | Two months
  We would like to know if the oncologists inform the patients the detailed management plan. and if they are expecting patients to fully understand the plan. This will be done via a questionnaire.
How satisfied do oncologists think most patients are during their management. | Two months
  we would like to know how satisfied are the patients during their management, and why they are unsatisfied from the oncologists point of view. This will be done via a questionnaire.
How often are Oncology patients open to their case being discussed in multidisciplinary clinics or being referred to psychiatrists/Nutritionists/palliative care/hospice? | Two months
  This will be done via a questionnaire to see their point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Riham AbdelAziz, MD/PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The questionnaire is aiming at exploring the thoughts and expectations of the medical staff in Oncology regarding their patients management and prognosis worldwide. It would be published after its completeion